CLINICAL TRIAL: NCT00731016
Title: Treatment of the Hutchinson-Gilford Progeria Syndrome With a Combination of Pravastatin and Zoledronic Acid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-002471-27; 2008-15
Record Dates: First submitted 2008-08-01; First posted 2008-08-08 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Hutchinson-Gilford Progeria Syndrome
MeSH Terms: conditions — Progeria | interventions — Zoledronic Acid; Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Zoledronic acid, pravastatin
  Interventions: Drug: Zoledronic acid, pravastatin

INTERVENTIONS:
Drug: Zoledronic acid, pravastatin — Pravastatin : 10 mg daily
  Zoledronic acid : slow (30 mn) intravenous injections, diluted into 50 ml of saline solution following this schedule :
  * injection 1, S1: 0.0125 mg/kg of zoledronic acid
  * injection 2, S6: 0.025 mg/kg of zoledronic acid
  * injection 3, S12 and following, trimestrial basis, 0.05 mg/kg of zoledronic acid

SUMMARY:
We suggest treating the Hutchinson-Gilford Progeria Syndrome by two molecules (zoledronic acid and pravastatin).The therapeutic approach which we propose has for objectives to reduce, to prevent or to delay the gravest infringements of the disease, to prolong the life of the children, and in a more general way, aim at improving their living conditions.

ELIGIBILITY:
Inclusion Criteria:

* Molecularly characterised patients with a known mutation of their LMNA gene leading to the production of a farnesylated prelamin A, whether truncated or not
* Patients must be able to travel and consult in Marseille, France for necessary explorations planned at the inclusion step, then following the protocol flow
* chart for zoledronic acid injections and follow-up visits
* Patient older than 3 years
* Patients affiliated or beneficiary of a legal medical insurance
* Adult patients certifying they have been properly informed about the protocol, and they signed a written consent form. Children and/or disabled patients whose parents/legal tutor have been informed and have signed a written consent form

Exclusion Criteria:

* Known hypersensitivity to pravastatin or zoledronic acid
* Seric transaminase levels higher than 3 times of normal value
* CPK level higher than 5 times of normal value
* Creatininemia higher than 0.5mg/dl or 44mM, or creatinin clearance lower than 70ml/min/1.73m3
* Presence of dental troubles, or recent dental trouble
* Maxillary osteonecrosis or bone nakedness antecedent
* Congenital galacosemia, glucose or galactose maladsorption syndrome, lactase deficiency
* Every other pathology thought to be incompatible with proposed treatment by the investigator
* Under treatment that can interfere with pravastatin and/or zoledronate metabolisms

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-10; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the tolerance and efficacy of pravastatin and zoledronic acid in combination on the patient's weight, height and bone metabolism in Progeria treatment | 48 months

SECONDARY OUTCOMES:
To evaluate the tolerance and efficacy of the treatment on other clinical and biological symptoms | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas LEVY, MD, Principal Investigator — Assistance Publique des Hopitaux de Marseille
Locations (1):
- Laboratoire de Génétique Moléculaire - Hopital de la Timone, Marseille, France